CLINICAL TRIAL: NCT03499145
Title: Validation of the Utility of Ophthalmology Intelligent Diagnostic System: A Clinical Trial
Brief Title: Validation of the Utility of Ophthalmology Intelligent Diagnostic System
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: Ministry of Health, China (Other Government); Xidian University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Clinical Professor, Sun Yat-sen University
Other Study IDs: CCPMOH2018-China-2
Record Dates: First submitted 2018-04-11; First posted 2018-04-17 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Ophthalmopathy; Artificial Intelligence
Keywords: conjunctivitis; keratitis; pterygium; cataracts
MeSH Terms: conditions — Eye Diseases; Conjunctivitis; Keratitis; Pterygium; Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Eligible patients for AI test.: Device: ophthalmology diagnostic system. An artificial intelligence to make comprehensive evaluation and treatment decision of ocular diseases.
  Interventions: Device: Ophthalmology diagnostic system.

INTERVENTIONS:
Device: Ophthalmology diagnostic system. — An artificial intelligence to make comprehensive evaluation and treatment decision of ocular diseases.

SUMMARY:
The prevention and treatment of diseases via artificial intelligence represents an ultimate goal in computational medicine. Application scenarios of the current medical algorithms are too simple to be generally applied to real-world complex clinical settings. Here, the investigators use "deep learning" and "visionome technique", an novel annotation method for artificial intelligence in medical, to create an automatic detection and classification system for four key clinical scenarios: 1) mass screening, 2) comprehensive clinical triage, 3) hyperfine diagnostic assessment, and 4) multi-path treatment planning. The investigator also establish a telemedicine system and conduct clinical trial and website-based study to validate its versatility.

ELIGIBILITY:
Inclusion Criteria:

* Patients and residents who underwent ophthalmic examination of the eye and recorded their ocular information in the outpatient clinic and community.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A prospective study of patients and residents who use the web platform for diagnosis.
Sampling Method: Probability Sample
Enrollment: 615 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
The proportion of accurate, mistaken and miss detection of the ophthalmology diagnostic system. | Up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Li W, Yang Y, Zhang K, Long E, He L, Zhang L, Zhu Y, Chen C, Liu Z, Wu X, Yun D, Lv J, Liu Y, Liu X, Lin H. Dense anatomical annotation of slit-lamp images improves the performance of deep learning for the diagnosis of ophthalmic disorders. Nat Biomed Eng. 2020 Aug;4(8):767-777. doi: 10.1038/s41551-020-0577-y. Epub 2020 Jun 22. PMID 32572198